CLINICAL TRIAL: NCT05861713
Title: Using Hydrating Cream to Improve Repeated Hand Skin Injury Among Tug-of-war Players: a Single Arm, Open-label, Split-hand Crossover Design Clinical Study
Brief Title: Using Hydrating Cream to Improve Repeated Hand Skin Injury Among Tug-of-war Players
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202300283A3
Record Dates: First submitted 2023-05-02; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Athletic Injuries; Eczematous Skin Diseases; Skin Avulsion
Keywords: Hydrating cream; Eczematous Skin Diseases; Skin Avulsion; Athletic Injuries
MeSH Terms: conditions — Athletic Injuries; Skin Diseases, Eczematous; Degloving Injuries

STUDY DESIGN:
Intervention Model Description: Evaluation of the efficacy of Hydrating Cream on Tug-of-war player with repeated hands injury by using a single arm, open-label, split-hand crossover design clinical study
Masking Description: Since the Hydrating Cream is applied to the subjects' hands and therefore masking is difficult to be done, the investigators adopt open-label design for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrating cream group (Experimental): The subjects will be instructed to apply the Hydrating Cream to the more severely affected side as the experimental group (e.g., the more severely injured left or right hand of tug-of-war athletes). At the same time, the other limb will be regarded as the control group. The study lasted for two weeks, and after two weeks, the experimental and control groups were switched, with the entire observation process lasting four weeks.
  Interventions: Drug: Hydrating Cream

INTERVENTIONS:
Drug: Hydrating Cream — The experimental group will apply the Hydrating Cream to the affected skin area at least twice daily with a cotton swab, while the other limb was the control group.

SUMMARY:
Athletes commonly face skin injuries during training and competition, which can negatively impact their performance and physical health. Injuries such as abrasions, cuts, burns, and sunburns can limit muscle contractions and range of motion, cause discomfort, and lead to bacterial infections. In addition, skin damage can lead to long-term skin problems such as skin aging and cancer, affecting athletes' overall health and performance. Protecting the skin is crucial for athletes to maintain optimal performance and physical health. The use of steroids is limited for athletes due to their status as banned substances. Topical steroids may also cause negative side effects, making it necessary to find alternative skin care options for athletes such as tug-of-war athletes. This study aims to evaluate the effectiveness of a topical hydrating cream for skin care in this population. The study involved using a moisturizing cream on the more severely affected side of one hand while the other hand acted as a comparative control group. After two weeks, the sides were switched, and the study continued for four weeks in total.

DETAILED DESCRIPTION:
Skin damage is a common issue for athletes. Whether during training or competition, athletes often face various skin injuries such as abrasions, cuts, bruises, burns, sunburns, etc. These injuries can have negative impacts on their body and performance, making the importance of protecting the skin self-evident. Firstly, skin damage may affect an athlete's sports performance. In an athlete's competition, any injury may affect their performance and result. Abrasions and bruises may limit muscle contractions, thereby affecting their ability and speed. Cuts and burns may also restrict their range of motion, especially in sports that require high flexibility, such as dance and gymnastics. Even minor injuries, such as blisters and abrasions, may cause discomfort and reduce their performance. Secondly, skin damage may also have negative impacts on an athlete's physical health. Abrasions and cuts may lead to bacterial infections, especially when using public facilities during competitions, such as showers and changing rooms. These infections may cause symptoms such as redness, fever, inflammation, and pus, and may require medication for treatment in severe cases. Sunburns and burns may lead to skin aging, skin cancer, and other skin problems, which may affect an athlete's long-term health and performance. Athletes have limited treatment options, as steroids are one of the important banned substances in sports. Even topical steroid creams may enter the bloodstream after long-term and widespread use, which can be detected in urine tests. Therefore, athletes should avoid using them as much as possible. In addition, topical steroids can cause side effects such as pigment deposition, skin thinning, bleeding, and even infection. Therefore, finding suitable topical medications for skin care in tug-of-war athletes is still necessary to avoid skin complications and potential impacts on performance. The purpose of this study is to clinically verify the effectiveness of the topical cream "Hydrating cream" for skin care in tug-of-war athletes and to evaluate its applicability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Dry and cracked skin lesions
* Not using any topical agents or emollients,

Exclusion Criteria:

* Malignancies or autoimmune disease-related skin lesions, such as psoriasis, systemic lupus erythematosus, dermatomyositis, etc.
* Under treatment of any kind or antibiotics
* Use oral, parental, or local corticosteroids in the recent one month
* Severe psychiatric illnesses, such as mania, major depression, bipolar or schizophrenia, etc.
* Known history of allergic to wool-related products.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in skin symptoms | day 0 (before use), day 14 (exchange date), and day 28 (end of the trial)
  The change in skin symptoms after using the Hydrating Cream will be evaluated using a visual analog scale, which ranges from 0 to 100, and a higher score indicates more severe skin symptoms.
Change in skin lesion area | day 0 (before use), day 14 (exchange date), and day 28 (end of the trial)
  The area of skin damage was estimated using the palmar method and recorded with photographs (excluding the face)

SECONDARY OUTCOMES:
Change in skin moisturization | day 0 (before use), day 14 (exchange date), and day 28 (end of the trial)
  Quantification of skin moisture. This will be assessed by GPskin Barrier Pro, which detects trans-epidermal water loss (TEWL) and stratum corneum hydration (SCH), both important indicators of skin moisturization.
Change in quality of life | day 0 (before use), day 14 (exchange date), and day 28 (end of the trial)
  Assessed using the generic EQ-5D-5L scale for overall quality of life and the Dermatology Life Quality Index (DLQI) for skin-related quality of life simultaneously

IPD SHARING:
Plan to Share IPD: No
The raw data sharing is only available on adequate request and could only be released if approved by the Institutional Review Board of the Chang Gung Medical Foundation.

REFERENCES:
- [Background] Hsieh CY, Tsai TF. Friction-Aggravated Skin Disorders-A Review of Mechanism and Related Diseases. Dermatitis. 2023 Jul-Aug;34(4):287-296. doi: 10.1097/DER.0000000000000961. Epub 2023 Jan 2. PMID 36255396
- [Background] McMullen E, Gawkrodger DJ. Physical friction is under-recognized as an irritant that can cause or contribute to contact dermatitis. Br J Dermatol. 2006 Jan;154(1):154-6. doi: 10.1111/j.1365-2133.2005.06957.x. PMID 16403110
- [Result] Logger JGM, Driessen RJB, de Jong EMGJ, van Erp PEJ. Value of GPSkin for the measurement of skin barrier impairment and for monitoring of rosacea treatment in daily practice. Skin Res Technol. 2021 Jan;27(1):15-23. doi: 10.1111/srt.12900. Epub 2020 Jun 23. PMID 32573826